CLINICAL TRIAL: NCT00418327
Title: Phase I Studies of TarcevaTM (Erlotinib Hydrochloride, OSI-774) as Single Agent in Children With Refractory and Relapsed Malignant Brain Tumors and in Combination With Irradiation in Newly Diagnosed Brain Stem Glioma
Brief Title: Safety Study of Tarceva in Children With Refractory and Relapsed Malignant Brain Tumors and Newly Diagnosed Brain Stem Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Geoerger Birgit/Coordinating Physician, Institut Gustave Roussy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSET 1120
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Malignant Brain Tumor; Brain Stem Glioma,
Keywords: Tarceva; refractory and relapsed malignant brain tumors; newly diagnosed brain stem glioma
MeSH Terms: conditions — Brain Neoplasms | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Tarceva (Erlotinib Hydrochloride) — tablets of 25 mg, 100 mg and 150 mg 75 to 150 mg/m² Once daily

SUMMARY:
The purpose of this study is to establish the recommended dose/Maximum Tolerated Dose (MTD) of Tarceva in children as single agent and in combination with radiation therapy

DETAILED DESCRIPTION:
Prognosis in relapsing malignant brain tumors is poor. Those in brain stem gliomas is dismal; median survival of these children does not exceed 9 months. Radiation therapy may result in early and transient amelioration of symptoms, but have not contributed to increase or prolong survival. Moreover, chemotherapy has not increased this outcome to date.Prados et al. reported encouraging results from a phase I study of TarcevaTM/OSI-774 alone or with temozolomide (TMZ) in patients with malignant gliomas. Of 25 evaluated patients, 6 experienced PR: 4 GBM (glioblastoma multiforme) and 1 grade 3 astrocytoma treated with TarcevaTM alone, 1 GBM treated with TarcevaTM/TMZ; 2 had minor responses, and 3 stable diseases. These results in malignant glioma and the lack of efficacy in brain stem glioma with current treatment suggests the evaluation of this new therapeutic agent in children with relapsed brain tumors and upfront at diagnosis in brain stem glioma in combination with radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant brain tumor
* Disease must be considered refractory to first line or relapsing after conventional therapy and for which no effective conventional treatment exists.·
* Newly diagnosed, histologically proven brain stem glioma, except pilocytic astrocytomas.
* Age: 1 to ≤ 21 years of age at study entry
* Life expectancy: at least 8 weeks
* ECOG Performance status ≤ 1 or Lansky-Play Scale>= 70%, and including children with motor paresis due to disease
* Measurable or evaluable disease
* No other serious concomitant illness
* No organ toxicity > grade 2 NCI-CTC AE v3.0, except alopecia and neurological symptoms due to disease

Exclusion Criteria:

* Patients with spontaneous intratumoral hemorrhage will not be included in the study, in exception of small post-biopsy hemorrhage due to biopsy procedure
* Pregnant and breast feeding woman
* Uncontrolled intercurrent illness or active infection
* Chemotherapy within 4 weeks prior to study medication (within 6 weeks, if the regimen contained a nitrosourea)
* Radiation therapy within 6 weeks prior to study medication
* Any clinical or non-clinical evidence of pulmonary dysfunction or pre-existing lung disease
* Severe cardiac pathology; history of myocardial infarction within the year prior to inclusion
* Any significant ophthalmologic abnormality, especially severe dry eye syndrome, keratoconjunctivitis sicca, Sjögren syndrome, severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions
* Treatment with Coumarin (warfarin)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-06

PRIMARY OUTCOMES:
To establish the recommended dose / Maximum Tolerated Dose (MTD) the for phase II study for single agent and in combination with radiation therapy | End of recruitment

SECONDARY OUTCOMES:
To define Dose Limiting Toxicities (DLTs) | 3 cycles-6 cycles
To define the safety profile | End of treatment
To characterize the pharmacokinetic behavior of TarcevaTM in children with brain tumors as a single agent and in combination with radiation therapy | Cycles 1,2,3,4,5,6
To evaluate efficacy | Cycles 2,4,6, end of treatment
To evaluate expression and mutations of EGFR with efficacy | End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vassal Gilles, Pr., Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] White-Koning M, Civade E, Geoerger B, Thomas F, Le Deley MC, Hennebelle I, Delord JP, Chatelut E, Vassal G. Population analysis of erlotinib in adults and children reveals pharmacokinetic characteristics as the main factor explaining tolerance particularities in children. Clin Cancer Res. 2011 Jul 15;17(14):4862-71. doi: 10.1158/1078-0432.CCR-10-3278. Epub 2011 Jun 8. PMID 21653689